CLINICAL TRIAL: NCT01977508
Title: The Vascutek Rapidax™ II Post Market Surveillance Registry
Status: Terminated | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: VAG-001
Record Dates: First submitted 2013-10-15; First posted 2013-11-06 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: End Stage Kidney Disease
Keywords: Vascular access grafts; Haemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- haemodialysis vascular access using ePTFE grafts
  Interventions: Device: ePTFE vascular access grafts

INTERVENTIONS:
Device: ePTFE vascular access grafts
  Other Names: RapidaxTM II Vascular access graft

SUMMARY:
Multicentre, prospective, observational post-market registry. To monitor and collect data on the post-market clinical safety and performance of the Vascutek Rapidax II Vascular Access Graft.

DETAILED DESCRIPTION:
At least 10 patients who have been implanted with a Rapidax II Vascular Access Graft for haemodialysis applications in patients with End Stage Renal Disease (ESRD), who are undergoing or are scheduled to begin haemodialysis and require implant of a prosthetic graft.

Primary End Points:Safety and Performance

* Secondary patency at 6 months post implant (Performance).(access survival until abandonment). The interval from time of implant to abandonment or time of measurement of patency, including intervention to re-establish the functionality of the thrombosed access
* Secondary patency at 12 months post implant (Performance.(access survival until abandonment). The interval from time of implant to abandonment or time of measurement of patency, including intervention to re-establish the functionality of the thrombosed access
* Freedom from device related Serious Adverse Events at 6 and 12 months (Safety)

Secondary End Points: Safety and performance

* Primary patency at 6 months post implant (Performance. (intervention free access survival). The interval from time of implant to any intervention designed to maintain or re-establish patency or to access thrombosis
* Primary patency at 12 months post implant (Performance).(intervention free access survival). The interval from time of implant to any intervention designed to maintain or re-establish patency or to access thrombosis
* Assisted primary patency at 6 months (Performance. (thrombosis free access survival). The interval from time of implant to intervention to maintain patency prior to the occurrence of thrombosis
* Freedom from device related Serious Adverse Events at 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 and ≤ 90 years old
2. Subject has a life expectancy of at least 12 months
3. Subject is scheduled to undergo placement of a new straight or loop arm arteriovenous haemodialysis access graft
4. The subject is willing and able to comply with the protocol and associated follow up requirements
5. Subjects must have agreed for their data to be entered into the registry as per the local hospital consent procedure

Exclusion Criteria:

1. Known allergy or sensitivity to ePTFE
2. Subject unwilling or unable to comply with the protocol
3. Life expectancy of less than 1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 10 patients who have been implanted with a Rapidax II Vascular Access Graft for haemodialysis applications in patients with End Stage Renal Disease (ESRD), who are undergoing or are scheduled to begin haemodialysis and require implant of a prosthetic graft.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety and Performance | 6 months
  * Secondary patency at 6 months post implant (Performance)
Safety and Performance | 12 months
  Secondary patency at 12 months post implant (Performance)
Safety and Performance | 12 months
  Freedom from device related Serious Adverse Events at 6 and 12 months (Safety)

SECONDARY OUTCOMES:
Safety and Performance | 6 months
  * Primary patency at 6 months post implant (Performance)
Safety and Performance | 12 months
  Primary patency at 12 months post implant (Performance)
  •
Safety and Performance | 12 months
  Assisted primary patency at 6 months (Performance)
  •
Safety and Performance | 12 months
  Freedom from device related Serious Adverse Events at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Lobenstein, Principal Investigator — Saale-Unstrut Klinikum Naumburg
Locations (3):
- Germany (3):
  - Saale-Unstrut Klinikum Naumburg, Naumburg
  - Thüringen Kliniken Georguis, Saale
  - Medinos Klinik Sonneberg, Sonneberg